CLINICAL TRIAL: NCT02717728
Title: Effectiveness of Fascia Iliaca Nerve Block for Post Hip Arthroscopy Pain Management: A Randomized Double-blind, Placebo Controlled Study
Brief Title: Effectiveness of Fascia Iliaca Nerve Block for Post Hip Arthroscopy
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: lack of funding
Sponsor: Boston Children's Hospital (Other)
Responsible Party: Principal Investigator, Karen Boretsky, Dr. Karen Boretsky, Boston Children's Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: IRB-P00021561
Record Dates: First submitted 2016-01-26; First posted 2016-03-24 (Estimated); Last update posted 2022-01-28 (Actual); Status verified 2022-01

CONDITIONS: Hip Surgery Corrective; Anesthesia; Functional

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Drug group Fascia iliaca nerve block (Active Comparator): Device: Fascia Iliaca Catheter placement Drug: Local anesthetic bolus :Ropivacaine 0.2% 0.5 ml/kg total in divided doses
  Device: Dressing: Catheter labeled: "Fascia Iliaca Catheter"
  Drug:Infusion: Ropivacaine 0.1%, rate: 0.3 ml/kg/hr; to start within the first hour after the block is placed. Infusion will be maintained for 24hs.
  Interventions: Procedure: Drug group Fascia iliaca nerve block
- Control group sham nerve block (Sham Comparator): Device: Fascia Iliaca Catheter placement (20 g catheter tip laid at appropriate insertion site)
  Device: Dressing: Catheter labeled: "Fascia Iliaca Catheter"
  Drug: Infusion: Ropivacaine 0.1% to plastic bag. rate: 0.3 ml/kg/hr; to start within the first hour after the block is placed. Infusion will be maintained for 24hs.
  Interventions: Procedure: Control group sham nerve block

INTERVENTIONS:
Procedure: Drug group Fascia iliaca nerve block — Device: Fascia Iliaca Catheter. Placement: Site prepared using aseptic technique.
  Device: Portable ultrasound: Localization of target site. Aseptic preparation of probe with sterile sheath. 18g x 10mm echogenic enhanced needle, 20G catheter inserted 3 cm beyond needle tip.
  Drug: Local anesthetic bolus: Ropivacaine 0.2% 0.5 ml/kg total in divided doses Device: Dressing Drug: Infusion of Ropivacaine 0.1%, rate: 0.3 ml/kg/hr; to start within the first hour after the block is placed. Infusion will be maintained for 24hs.
  Arms: Drug group Fascia iliaca nerve block
Procedure: Control group sham nerve block — Device: Fascia Iliaca Catheter placement: Site prepared using aseptic technique.
  Device: portable ultrasound: Localization of target site. Aseptic preparation of probe with sterile sheath.
  Device: Dressing
  Drug: Infusion of Ropivacaine 0.1%, rate: 0.3 ml/kg/hr; to start within the first hour after the block is placed. Infusion will be maintained for 24hs.
  Arms: Control group sham nerve block

SUMMARY:
There is currently no standard of care or best practice for managing post-operative pain for patients undergoing hip arthroscopy. Perioperative pain with these procedures can be substantial. It has been shown that up to 90% of patients in the Post-anesthesia care unit (PACU) following hip arthroscopy report pain scores of 7/10. Poor pain management following hip fracture surgery directly results in increased time spent in high cost health care areas and delayed time to ambulation. Continuous regional anesthesia following hip arthroplasty has been shown to reduce narcotic consumption and related side-effects (reduction of post-operative pain, delirium, and length of stay).

The purpose of this research is to evaluate the effectiveness of a fascia iliaca nerve block in reducing post-operative pain within the first 24 hours following hip arthroscopy. Additionally, the pharmacokinetics of the drug ropivacaine will be studied via laboratory analysis of blood samples. Ultimately, the objective of this research is to develop a standard of care or best practice for the management of post-operative pain following hip arthroscopy. This study will include the entire age range of patients who are seen for hip arthroscopy at Boston Children's Hospital, for which there is a 35 year age limit. Both sexes will be included in the study.

The study design will be real catheter versus a sham catheter(control). All subjects will receive general anesthesia. The catheters (real or sham) will be administered after the induction of general anesthesia and before the beginning of the surgery until 24 hours after recorded PACU admittance time. The anesthesia team placing the block will not be blinded. The orthopaedic surgeon (Dr. Yen) and all evaluators will be blinded to the absence or presence of a real catheter. In the case of a sham catheter, the anesthesia team will rig a pump to look like it is dispensing local anesthesia.

To determine the pharmacokinetics of ropivicaine during standard fascia iliaca block, following induction of general anesthesia, a large bore IV catheter will be inserted for the purpose of blood draws (all patients).

DETAILED DESCRIPTION:
This study will be a randomized, double-blinded, placebo controlled study. All patients who are scheduled to undergo a hip arthroscopy with Dr. Yen who meet the inclusion/exclusion criteria will be approached and informed consent and assent when indicated would be obtained.Attending surgeon, anesthesia care team, PACU nursing staff, inpatient ward nursing staff and evaluators will be blinded to study group. Regional Anesthesia team and pharmacy staff will be not blinded to assignment of patient group but will have no additional contact with patient after provision of sham or actual perineural catheter. the study design will be real catheter versus a sham catheter, or control. All subjects will receive general anesthesia. The catheters (real or sham) will be administered after the induction of general anesthesia and before the beginning of the surgery until 24 hours after recorded PACU admittance time. The anesthesia team placing the block will not be blinded. The orthopaedic surgeon (Dr. Yen) and all evaluators will be blinded to the absence or presence of a real catheter. In the case of a sham catheter, the anesthesia team will rig a pump to look like it is dispensing local anesthesia.

1. General Anesthesia a) Induction (IV): i. propofol: 2-4 mg/kg [9] ii. fentanyl: 2 mcg/kg administered iii. decadron: 4 mg as an antiemetic b) Airway: i. Airway management will be chosen by the anesthesiologist in charge of the case.

   c) Maintenance of anesthesia i. Sevoflurane 1.1 minimum alveolar concentration (MAC) ii. If heart rate or blood pressure increase > 20% above baseline (tachycardia as determined the morning of surgery in the holding area), anesthesiologist will administer1 microgram/kg fentanyl as bolus. May repeat as often as every 10 minutes. Maximum 8 doses.

   iii. With patient movement, anesthesiologist will administer propofol 1 mg/kg intravenous push. May repeat every 5 minutes as necessary.

   d) Emergence i. Discontinue isoflurane ii. Zofran 4 mg IV iii. Ketorolac 0.5 mg/kg IV; max dose 30 mg.
2. Perineural Catheter:

   * Actual and sham will be hooked to infusion pump and receptacle
   * Pharmacy will label the infusion pumps, and will cover these labels in such a way that the cover can be immediately at any point if needed.
   * Regional anesthesia team will double check the correct direction of the stopcock of the tubing set.

     a) Drug Group: i. Fascia Iliaca Catheter placement
     1. Administrator: Regional Anesthesiologist

        1. Minimum of three years anesthesia training
        2. Cannot be blinded, but will not contact/communicate with patient after surgery
     2. Appropriate laterality identified
     3. Site prepared using aseptic technique
     4. Localization of target site beneath fascia iliaca plane using portable ultrasound

        1. Aseptic preparation of probe with sterile sheath
        2. 38mm linear probe (BK Medical, USA)
        3. 15 MHz frequency
     5. Needle: 18g x 10mm echogenic enhanced needle
     6. 20G catheter inserted 3 cm beyond needle tip ii. Local anesthetic bolus

     <!-- -->

     1. Ropivacaine 0.5 ml/kg total in divided doses

        a. Aspirate every 5 ml
     2. Administered via needle iii. Dressing:

     1. Liquid adhesive to skin 2. Sorbaview dressing (2x2) applied directly over catheter on skin 3. Catheter coiled once on top sorbaview and clear plastic dressing applied over sorbaview 4. 3x3 gauze taped over dressing to cover insertion site 5. Catheter labeled: "Fascia Iliaca Catheter" b) Control Group i. Fascia Iliaca Catheter placement

     1. Administrator: Regional Anesthesiologist
     1. Minimum of three years anesthesia training
     2. Cannot be blinded, but will not contact/communicate with patient after surgery 2. Appropriate laterality of surgery identified 3. Site prepared using aseptic technique 4. Localization of target site beneath fascia iliaca plane using portable ultrasound

     a. Aseptic preparation of probe with sterile sheath b. 38mm linear probe (BK Medical, USA) c. 15 MHz frequency 5. 20 g catheter tip laid at appropriate insertion site ii. Dressing:

     1. Liquid adhesive to skin 2. Sorbaview dressing (2x2) applied directly over catheter on skin 3. Catheter coiled once on top sorbaview and clear plastic dressing applied over sorbaview 4. 3x3 gauze taped over dressing to hide insertion site 5. Catheter labeled: "Fascia Iliaca Catheter"
3. Infusion

   a) Pharmacy to prepare and label all infusion syringes b) Actual content (ropivacaine 0.1%) to be covered but immediately available in case of need to know. Violation of blinding to be obvious when tubing set removed. A non-blinded member of the study team will remove the set.

   i. Drug Group: Ropivacaine 0.1% ii. Control: Ropivacaine 0.1% to plastic bag c) Device: bodyguard infusion pump d) Rate: 0.3 ml/kg/hr; max 15 to start within the first hour after the block is placed.

   e) Infusion bag to be changed out as needed by nursing staff per usual routine (depends on volume of bag, weight of patient)
4. Surgical Procedure

   1. Hip arthroscopy performed i. Pre-operative:

      1. Patient padded, per usual method
      2. Range Of Motion check by Yen and/or surgical staff
      3. Patient placed in traction device
      4. Xrays taken (AP pelvis, Dunn, frog leg, false profile). Must get view of lesion.
      5. Leg prepped/draped in normal fashion
   2. At conclusion of surgical procedure, patients in both groups to receive standard local anesthetic infiltration i. 20 cc total

      1. 10 ml 0.2% ropivacaine intra-articular into hip joint
      2. 5 ml 0.2% ropivacaine to each trochlear site (x2) Post-operative Methods

   All patients will remain in the hospital for a minimum of 24 hours following surgery per Dr. Yen's normal hip arthroscopy standard of care. A blinded observer will record pain scores at 30 minutes, 1 hour, 2 hours, 4 hours, 6 hours, and 24 hours postoperatively. Pain scores will be measures at rest by an 11-point numeric rating scale (NRS) ranging from 0-10, where 0 is no pain and 10 is worst pain imaginable. All patients should complete the study and have measurements at each time point. Patient demographics including age and gender as well as surgical characteristics including length of surgery, estimated blood loss, and surgery type will be recorded.

   Blinded observers will also record the time until patients require additional morphine, the amount of morphine consumed at each time it was requested, and whether the patient reported nausea or experienced vomiting within the first 24 hours post-operatively.
5. PACU a) Time 0 = PACU arrival time b) Pain scores: i. Obtained by trained, blinded nurse observers ii. Recorded per policy with minimum evaluation every 15 minutes iii. Recorded using 11 point numeric rating scale (NRS) 1. 0 = no pain; 10 = severe pain c) PCA (patient controlled analgesia) available and initiated upon arrival to PACU i. Opioid: morphine ii. Bolus dose: 0.025 mg/kg; lockout 10 minutes iii. Hourly limit: 0.15 mg/kg/hr iv. Nurse rescue bolus: 0.05 mg/kg; lockout 60 minutes 1. To be administered for NRS > 7 v. continuous hourly infusion = 0
6. Inpatient Wards

   1. Nurses will evaluate pain per usual practice. Documented minimum every 4 hours. i. pain scores >7, nurse will administer: nurse rescue bolus via PCA ii. No dermatome test to prevent the introduction of bias by inadvertently un-blinding subjects.

Pharmacokinetic Methods To determine the pharmacokinetics of ropivicaine during standard fascia iliaca block [10-13].

1. Following induction of general anesthesia, a large bore IV catheter will be inserted for the purpose of blood draws (all patients)
2. Blood Sampling (all patients)

   1. Volume 2ml
   2. Time = zero defined as immediately following bolus of ropivicaine or sham equivalent
   3. First hour: collected at 5, 10, 15, 30, 35, and 60 minutes.
3. Analysis:

   1. Internal lab
   2. Blood samples will be centrifuged to separate the plasma and stored at -20 degrees C until assay. Plasma ropivacaine levels analyzed by gas chromatography

ELIGIBILITY:
Inclusion Criteria:

1. Patient age at surgery is 12-35.
2. Able to provide informed consent and/or assent.
3. Diagnosis is Femoro-acetabular impingement (FAI) and/or labral tear.
4. Surgery will involve and be limited to hip arthroscopy and osteoplasty of the acetabular rim or femoral head/neck junction.
5. Surgery will be performed by Dr. Yi-Meng Yen.
6. Admission status: 24 hour admission to hospital.
7. No contraindication to study procedures

Exclusion Criteria:

1. Hip revision surgery
2. Underlying neurologic disorder affecting pain perception.
3. Underlying neurocognitive disorder or developmental delay affecting ability to convey feelings of pain to medical staff.
4. Underlying opioid use or addiction.
5. Significant concomitant hip pathology.
6. Active infection over catheter site.
7. History of chronic pain (not localized to the hip) requiring consistent opioid consumption for greater than or equal to 6 months within year prior to surgery.
8. Allergy to local anesthetics
9. Allergy to fentanyl
10. Allergy to midazolam
11. Allergy to morphine
12. American Society of Anesthesia class 3 or higher.

Ages: 12 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 0 (Actual)
Dates: Start 2020-12 (Estimated); Primary Completion 2021-12 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
The investigators will measure morphine consumption as the endpoint, to compare the efficacy of each group | Within the first 24hs after the fascia iliaca block is placed.

SECONDARY OUTCOMES:
The investigators will collect postoperative pain scores using the 11 point numeric rating scale in each group, to compare the efficacy of each group | Within the first 24hs after the fascia iliaca block is placed.
The investigators will collect time to first opioid consumption in each group, To compare the efficacy of each group. | Within the first 24hs after the fascia iliaca block is placed.
The investigators will document incidence of postoperative nausea and vomiting in each group. | Within the first 24hs after the fascia iliaca block is placed.
The investigators will measure maximum plasma concentrations at specific time intervals of 0.2% ropivacaine administered via a fascia iliaca block. | Within the first hour after the fascia iliaca block is placed.

CONTACTS AND LOCATIONS:
Overall Officials: Yi-Meng Yen, MD, Principal Investigator — Boston Children's Hospital
Locations (1):
- Boston Children's Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Paut O, Schreiber E, Lacroix F, Meyrieux V, Simon N, Lavrut T, Camboulives J, Bruguerolle B. High plasma ropivacaine concentrations after fascia iliaca compartment block in children. Br J Anaesth. 2004 Mar;92(3):416-8. doi: 10.1093/bja/aeh066. Epub 2004 Jan 22. PMID 14742340
- [Result] Ward JP, Albert DB, Altman R, Goldstein RY, Cuff G, Youm T. Are femoral nerve blocks effective for early postoperative pain management after hip arthroscopy? Arthroscopy. 2012 Aug;28(8):1064-9. doi: 10.1016/j.arthro.2012.01.003. Epub 2012 Apr 11. PMID 22498045
- [Result] Morrison SR, Magaziner J, McLaughlin MA, Orosz G, Silberzweig SB, Koval KJ, Siu AL. The impact of post-operative pain on outcomes following hip fracture. Pain. 2003 Jun;103(3):303-311. doi: 10.1016/S0304-3959(02)00458-X. PMID 12791436
- [Result] Smith HS, Laufer A. Opioid induced nausea and vomiting. Eur J Pharmacol. 2014 Jan 5;722:67-78. doi: 10.1016/j.ejphar.2013.09.074. Epub 2013 Oct 21. PMID 24157979
- [Result] Marino J, Russo J, Kenny M, Herenstein R, Livote E, Chelly JE. Continuous lumbar plexus block for postoperative pain control after total hip arthroplasty. A randomized controlled trial. J Bone Joint Surg Am. 2009 Jan;91(1):29-37. doi: 10.2106/JBJS.H.00079. PMID 19122076
- [Result] Rashiq S, Vandermeer B, Abou-Setta AM, Beaupre LA, Jones CA, Dryden DM. Efficacy of supplemental peripheral nerve blockade for hip fracture surgery: multiple treatment comparison. Can J Anaesth. 2013 Mar;60(3):230-43. doi: 10.1007/s12630-012-9880-8. Epub 2013 Jan 19. PMID 23334780